

# **Trial Statistical Analysis Plan**

c17305575-01

**BI Trial No.:** 1386.8

**Title:** Safety, tolerability, pharmacokinetics and pharmacodynamics of

multiple rising oral doses of BI 1467335 in healthy male and female subjects (double-blind, randomised, placebo-controlled

within dose groups)

(Including protocol amendment 1 (c08854973-02), amendment 2

(c08854973-03) and amendment 3 (c08854973-04))

**Investigational** 

**Product:** 

BI 1467335

Responsible trial statisticians:

Phone:

Fax:

Phone: Fax:

Date of statistical analysis plan:

29 Aug 2017 SIGNED

Version:

Final

**** 

Proprietary confidential information

© 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

#### **TABLE OF CONTENTS** 1.

| TITLE | PAGE | 1 |
|--------------|------------------------------------------------|-----------|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINT | |
| 5.2.1 | Key secondary endpoint | |
| 5.2.2 | Secondary endpoint | |
| 5.3.2 | Safety parameters | 10 |
| | Salet, parameters | 10 |
| 6. | GENERAL ANALYSIS DEFINITIONS | 14 |
| 6.1 | TREATMENTS | |
| 6.2 | IMPORTANT PROTOCOL VIOLATIONS | |
| 6.3 | SUBJECT SETS ANALYSED | |
| 6.3 | | |
| 6.5 | POOLING OF CENTRES | 17 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 17 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 18 |
| 7. | PLANNED ANALYSIS | 21 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 21 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 22 |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINTS | 22 |
| 7.5 | SECONDARY ENDPOINT | 22 |
| 7.5.1 | Key secondary endpoint | 22 |
| 7.5.2 | Secondary endpoints | 22 |
| <b>7.6.2</b> | Safety parameters | <u>23</u> |
| 7.7 | EXTENT OF EXPOSURE | 24 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| <b>7.8</b> | SAFETY ANALYSIS | 25 |
|--------------|----------------------------------------------------|------|
| <b>7.8.1</b> | Adverse events | . 25 |
| <b>7.8.2</b> | Laboratory data | .26 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | .27 |
| 7.8.5 | Others | . 29 |
| 8. | REFERENCES | .30 |
| 9. | ADDITIONAL SECTIONS | .31 |
| 9.1 | DETAILED DESCRIPTION OF ENDPOINTS FOR ECG | .31 |
| 9.2 | STEPS IN CASE OF CONVERGENCE PROBLEMS FOR REPEATED | |
| | MEASURES MODEL IN ECG | .32 |
| 10. | HISTORY TABLE | .34 |

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Flow chart of analysis phases for statistical analyses of AEs, safety | |
|---|---|---|
| | laboratory data, vital signs and ECG | 14 |
| Table 6.2: 1 | Important protocol violations | 15 |
| Table 6.3: 1 | Subject sets analysed | 17 |
| Table 6.7: 1 | Time schedule of 12-lead ECG recordings | 18 |
| Table 10: 1 | History table | 34 |

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADME | Absorption, distribution, metabolism, and excretion |
| ADS | Analysis dataset |
| AE | Adverse event |
| Ae <sub>0-24,N</sub> | Amount of analyte eliminated in urine over 24 h after administration of the $N^{\rm th}$ dose |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUC <sub>0-24</sub> | Area under the concentration-time curve of the analyte in plasma over<br>the time interval from 0 to 24 hours after administration of the first<br>dose |
| AUC <sub>0-24,28</sub> | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours after administration of the 28 <sup>th</sup> dose |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BMI | Body mass index |
| BMS | Biomarker set |
| $C_{1,N}$ | Concentration of the analyte in plasma 1 hour after administration of the $N^{\rm th}$ dose |
| CARE | Clinical data analysis and reporting environment |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma after administration of the first dose |
| $C_{\text{max},28}$ | Maximum measured concentration of the analyte in plasma following administration of the 28 <sup>th</sup> dose |
| $C_{\text{pre},N}$ | Predose concentration of the analyte in plasma immediately before administration of the $N^{\text{th}}$ dose after $N$ - $I$ doses were administered |
| CRF | Case report form |
| CTCAE | Common terminology criteria for adverse events |
| CTP | Clinical trial protocol |
| CTR | Clinical trial report |
| CV | Arithmetic coefficient of variation |
| DBLM | Database lock meeting |

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| DNA | Deoxyribonucleic acid |
| ECG | Electrocardiogram |
| ECGPCS | Electrocardiogram plasma concentration set |
| eCRF | Electronic case report form |
| EMA | European Medicines Agency |
| EudraCT | European union drug regulating authorities clinical trials |
| gCV | Geometric coefficient of variation |
| gMean | Geometric mean |
| HR | Heart rate |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| IPV | Important protocol violation |
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NOA | Not analysed |
| NOR | No valid result |
| NOS | No sample available |
| on-trt | on-treatment |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| PKS | Pharmacokinetic parameter analysis set |
| PR interval | ECG interval from the onset of P wave to the beginning of the QRS |
| PV | Protocol violation |
| QRS complex | Combination of the Q, R, and S waves |
| QT interval | ECG interval from the beginning of the QRS complex to the end of the T wave |
| QTcB | QT interval, heart rate corrected according to Bazett's formula |
| QTcF | QT interval, heart rate corrected according to Fridericia's formula |
| QTcN | QT interval, heart rate corrected according to study population formula |
| R | Reference treatment |
| RAGe | Report appendix generator |
| RPM | Report planning meeting |
| RR interval | ECG interval from the peak of the R wave to the peak of the subsequent R wave |

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Тоши | Definition / description |
|------|---------------------------------|
| Term | Definition / description |
| RS | Randomised set |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SDL | Subject data listing |
| SOC | System organ class |
| T | Test treatment |
| TS | Treated set |
| TSAP | Trial statistical analysis plan |
| ULN | Upper limit of normal range |

#### 3. INTRODUCTION

As per ICH E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle Clinical<sup>TM</sup> system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.



QTcN correction was added as additional further ECG parameter to be evaluated.

### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

Primary endpoint is the number [N (%)] of subjects with drug-related AEs, as defined in Section 5.2.1 of the CTP.

#### 5.2 SECONDARY ENDPOINT

### 5.2.1 Key secondary endpoint

Not applicable.

### **5.2.2** Secondary endpoint

Secondary endpoints are  $AUC_{0-24}$ ,  $C_{max}$ ,  $AUC_{0-24,28}$  and  $C_{max,28}$  of BI 1467335 in plasma, as defined in Section 5.5.1.1 of the CTP.



### 5.3.2 Safety parameters

**CTP:** Further criteria of interest:

- AEs (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (blood pressure, pulse rate)
- Exclusion of cataract formation

#### 12-lead ECG endpoints

For the definition of baseline and a summary of time points please refer to Section 6.7.

#### **Quantitative ECG endpoints:**

The following quantitative ECG endpoints will be determined for the ECG variables QTcN, QTcF, QT, HR, PR, QRS, RR and QTcB derived as described in Additional Section 9.1:

- absolute values (per time point)
- changes from baseline (per time point)
- percent changes from baseline (per time point; for HR, PR, QRS)

### Categorical ECG endpoints

The following categorical ECG endpoints will be determined based on the quantitative ECG endpoints:

- New onset (meaning that this or a higher category was not present at baseline) of maximum QTcN interval > 450 to 480 msec, > 480 to 500 msec, or > 500 msec on treatment (and similar for QTcF).
  For assignment of a particular subject to one of the above categories, all time points ontreatment (refer to Table 6.7: 1) will be considered. If baseline is missing, but the maximum absolute QTcN interval falls in a category other than normal (i.e. when QTcN > 450 msec), then this is categorized as a new onset in the respective category. If baseline is missing, but the maximum absolute QTcN interval is normal, then it is categorized as "No new onset" (similar for QTcF).
- Maximum change from baseline in QT interval  $\leq$  60 msec, or > 60 msec on treatment
- Maximum change from baseline in QTcN interval  $\leq 30$  msec, > 30 to  $\leq 60$  msec, or > 60 msec on treatment (similar for QTcF)

The occurrence of any of the following will be viewed as "notable findings":

- New onset (not present at baseline) of uncorrected QT interval > 500 msec at any time on treatment
  - If baseline is missing, any occurrence of QT interval > 500 msec at any time on treatment will be a notable finding
- New onset of QTcN interval > 500 msec at any time on treatment (and similar for QTcF) If baseline is missing, any occurrence of QTcN interval > 500 msec at any time on treatment will be a notable finding (similar for QTcF)
- Increase in QTcN interval from baseline by > 60 msec at any time on treatment (similar for QTcF)
- Increase in HR from baseline by  $\geq 25\%$ , when corresponding on-treatment value of HR is > 100 beats/min, or decrease in HR by  $\geq 25\%$ , when corresponding on-treatment value of HR is < 50 beats/min, at any time on treatment
- Increase in the PR interval from baseline by  $\geq 25\%$ , when corresponding on-treatment value of PR interval is > 200 msec, at any time on treatment
- Increase in the QRS complex from baseline by  $\geq 10\%$ , when corresponding on-treatment value of QRS complex is > 110 msec, at any time on treatment

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignments of dose groups, and selection of doses, cf. Section 4 of the CTP.

Subjects will be treated with 10 mg, 15 mg or 20 mg of BI 1467335 (test treatment, T) or placebo (reference treatment, R) once daily over 28 days. All placebo subjects will be analysed in one pooled placebo group (i.e. no distinction between dose groups will be made for placebo subjects).

For statistical analysis of AEs, safety laboratory data, vital signs and ECG, the following analysis phases are defined for each subject:

Table 6.1: 1 Flow chart of analysis phases for statistical analyses of AEs, safety laboratory data, vital signs and ECG

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening | Screening | Date of informed consent | Date/time of first administration of study drug |
| On-treatment | Placebo,<br>10 mg BI,<br>15 mg BI,<br>or 20 mg BI,<br>respectively | Date/time of first administration of study drug | 12:00 AM on day after<br>subject's trial termination<br>date |

CTR Section 15, Appendix 16.1.9.2.8.2 and Appendix 16.1.9.2.8.3 AE displays will present results for the on-treatment phase only.

In CTR Section 15 AE tables (but not in Appendix 16.1.9.2.8.2 and Appendix 16.1.9.2.8.3 AE tables), the following totals will be provided in addition:

- "Total BI", defined as the total over all on-treatment phases involving BI, i.e., "10 mg BI" + "15 mg BI" + "20 mg BI"
- "Total on-trt", defined as the total over all on-treatment phases, i.e., "Placebo" + "10 mg BI" + "15 mg BI" + "20 mg BI"

CTR Appendix 16.1.9.2.8.1 displays will present results for the screening and on-treatment phases.

Additionally to the totals defined above, the following total will be provided in CTR Section 16.1.9.2.8.1 AE tables:

• "Total", defined as the total over all study phases (screening + on-treatment)

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL VIOLATIONS

Consistency check listings (for identification of violations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the RPM/DBLM. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an IPV. For definition of IPVs, and for the process of identification of these, refer to the BI reference document "Protocol Violation Handling Definitions" (1).

If any IPVs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet (2). The following table contains the categories which are considered to be IPVs in this trial. If the data show other IPVs, this table will be supplemented accordingly by the time of the RPM/DBLM.

IPVs will be summarised and listed.

Table 6.2: 1 Important protocol violations

| Cate | egory<br>ode | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C2 | Randomisation not followed |
| | C3 | Non-compliance |
| | C4 | Medication code broken inappropriately |
| | C5 | Incorrect intake of trial medication |
| D | | Concomitant medication |
| | D1 | Prohibited medication use |
| E | | Missing data |
| | | Certain violations of procedures used to measure primary or secondary data |

Violations C1, C2, C4, and C5 can only be detected at the trial site.

Source: BI reference document "Protocol Violation Handling Definitions" [001-MCS-50-413 RD-01] (1).

#### 6.3 SUBJECT SETS ANALYSED

The following subject sets will be defined for statistical analysis:

- Randomised set (RS): This subject set includes all subjects who were randomised, i.e., who have been assigned a subject number, whether treated or not.
- Treated set (TS):
  This subject set includes all subjects who received at least one dose of study drug, as defined in Section 7.3.1 of the CTP. This is the full analysis set population in the sense of ICH-E9.
- Pharmacokinetic parameter analysis set (PKS):
  This subject set includes all subjects of the TS who provide at least one PK parameter that was not excluded due to relevant PVs or due to PK non-evaluability, as defined in Section 7.3.1 of the CTP.



All ECG analyses are performed on the TS, except for the exposure-response analyses, which are performed on the ECGPCS defined below.

• ECG PC set (ECGPCS):

This subject set consists of all subjects in the TS who provide a baseline value and at least one post-baseline value for at least one ECG variable used in the exposure-response analysis, and a corresponding (i.e. time-matched) valid drug plasma concentration. Since placebo subjects will be included in the exposure-response analyses with plasma concentration set to 0, a plasma concentration BLQ is considered a valid drug plasma concentration for placebo subjects.

The discussion of all exceptional cases and problems and the decisions on the allocation of subjects to analysis sets will be made at latest at the RPM/DBLM.

Table 6.3: 1 Subject sets analysed

| | | | Subject set | : | |
|---|---|---|---|---|---|
| Class of endpoint | RS | TS | PKS | BMS | ECGPCS |
| Disposition | X | X | | | |
| Exposure | | X | | | |
| IPVs | X | | | | |
| Demographic/baseline endpoints | | X | | | |
| Primary endpoint | | X | | | |
| ECG endpoints and plasma concentrations used in exposure-response analysis | | | | | X |
| ECG endpoints in other analyses | | X | | | |
| Other safety parameters | | X | | | |
| Secondary PK endpoints | | | X | | |



#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

**CTP**: If a subject is removed from or withdraws from the trial prior to first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) or trial database and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In this case, the data will be included in the CRF/trial database and will be reported in the CTR.

**CTP**: With respect to safety evaluations, it is not planned to impute missing values.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156\_RD-01 (3)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472\_RD-01) (4). CTP: For tabulation and graphical displays, drug concentration data identified with NOS (no sample available), NOR (no valid result), NOA (not analysed), or

BLQ (below the lower limit of quantification) will be displayed as such and not replaced by zero at any time point (this rule also applies also to the lag phase, including the predose values).

**CTP**: For the calculation of PK parameters by non-compartmental analysis, concentration data identified with NOS, NOR or NOA will generally not be considered. Concentration values in the lag phase identified as BLQ will be set to zero. All other BLQ values of the profile will be ignored. The lag phase is defined as the period between time zero and the first time point with a concentration above the quantification limit.

**CTP**: *No imputation of missing PK parameters will be performed.* 



#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

There will be a centralised evaluation of all 12-lead ECG recordings at the time points specified in Table 6.7: 1 below:

Table 6.7: 1 Time schedule of 12-lead ECG recordings

| Visit | Day | Planned time [hh:mm] (relative to drug administration) | Study phase |
|---|---|---|---|
| 2 | 1 | -02:00 | Baseline |
| | | 00:15 | On-treatment |
| | | 00:30 | |
| | | 00:45 | |
| | | 01:00 | |
| | | 01:30 | |
| | | 02:00 | |
| | | 04:00 | |
| | | 08:00 | |
| | | 12:00 | _ |
| | 2 | 24:00 | |
| | 3 | 48:00 | |
| | 4 | 72:00 | |
| | | 73:00 | |

Table 6.7: 1 Time schedule of 12-lead ECG recordings (continued)

| Visit | Day | Planned time | Study phase |
|-------|-----|--------------|-------------|
|-------|-----|--------------|-------------|

| | | [hh:mm] | |
|---|----|-----------------------------------|--------------|
| | | (relative to drug administration) | |
| 2 | 7 | 144:00 | On-treatment |
| 2 | | | On-treatment |
| | 14 | 145:00 | |
| | 14 | 310:00 | - |
| | | 312:15 | _ |
| | | 312:30 | 4 |
| | | 312:45 | _ |
| | | 313:00 | _ |
| | | 313:30 | 4 |
| | | 314:00 | _ |
| | | 316:00 | |
| | | 320:00 | |
| | | 324:00 | |
| | 15 | 336:00 | |
| | 16 | 360:00 | |
| | 17 | 384:00 | |
| | | 385:00 | |
| | 21 | 480:00 | |
| | | 481:00 | |
| | 28 | 646:00 | |
| | | 648:15 | |
| | | 648:30 | |
| | | 648:45 | 7 |
| | | 649:00 | 7 |
| | | 649:30 | |
| | | 650:00 | |
| | | 652:00 | 7 |
| | | 656:00 | 7 |
| | | 660:00 | 7 |
| | 29 | 672:00 | 7 |

Triple ECGs (3 single ECGs recorded within 180 sec) will be recorded on all time points on Day 1, Day 2, Day 14, Day 15, Day 21, Day 28 and Day 29. On all other time points, single ECGs will be recorded.

The value of an ECG variable at each of the time points with triple ECG is defined as the arithmetic mean of the 3 single ECG measurements. In particular, the baseline value of an

ECG variable is defined as the mean of the triple ECG measurements prior to first drug administration.

In all other analyses (except for analyses of ECG variables), the last non-missing value determined prior to the first dosing of BI 1467335 will be defined as baseline.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM/DBLM.

### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (001-MCG-159) (9).

The individual values of all subjects will be listed. Listings will generally be sorted by dose group, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

Inferential statistical analyses of secondary and further PK endpoints will be performed by and will be presented in Section 15.5 of the CTR and in Appendix 16.1.9.3

Descriptive data analysis of PK will be performed by BI and presented in Sections 15.6 and 15.7 of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters and biomarker parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary.

Only descriptive statistics are planned for this section of the CTR.

A medication will be considered concomitant to a treatment, if it

- is ongoing at the time of first administration of the respective treatment or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Refer to Section 7.8.1 for a description of the analysis of AEs, and in particular the analysis of the frequency of subjects with drug related AEs, which is the primary endpoint of this trial.

#### 7.5 SECONDARY ENDPOINT

#### 7.5.1 Key secondary endpoint

Not applicable.

#### 7.5.2 Secondary endpoints

The analysis of secondary endpoints will be based on the PKS.

Dose proportionality of secondary endpoints will be evaluated as defined in the CTP, Section 7.3.1, by use of the power model. If steady state will already be reached after 14 days of treatment, dose proportionality will also be investigated for  $AUC_{0-24,14}$  and  $AUC_{0-24,28}$  together (and for  $C_{max,14}$  and  $C_{max,28}$  together, respectively) by use of a repeated measurements model, as described in Section 7.3.1 of the CTP.

#### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

#### Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (5).



#### 7.6.2 Safety parameters

Safety and tolerability will be analysed as described in <u>Section 7.8</u> of this TSAP.



TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 7.7 **EXTENT OF EXPOSURE**

Only descriptive statistics are planned for this section of the CTR.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity [CTCAE grade Version 4.03], action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Handling and summarization of adverse event data for clinical trial reports and integrated summaries" (6) [001-MCG-156] and "Handling of missing and incomplete AE dates" (3) [001-MCG-156\_RD-01].

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to the screening phase or on-treatment phase as defined in Section 6.1.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 and for the class of AESIs.

**CTP:** The following are considered as AESIs in this trial:

- Hepatic injury, as defined by the following alterations of hepatic laboratory parameters:
  - o an elevation of AST and/or ALT  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, and/or
  - $\circ$  marked peak aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN.

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (8), AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or
- (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related (primary endpoint) will be summarised separately. Separate tables will also be provided for subjects

with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (8)). The frequency of subjects with AEs and the frequency of subjects with AEs considered by the investigator to be drug related will also be summarised by maximum grade of CTCAE (version 4.03), primary SOC and preferred term.

The SOCs will be sorted according to the standard sort order specified by the EMA, preferred terms will be sorted by total frequency (within SOC).

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (7). Due to inclusion of male and female subjects, laboratory analyses will be based on normalised values, i.e., for a given laboratory parameter, values will be transformed to a standard unit and a standard reference range before statistical analysis.

**CTP:** Laboratory data will be compared to their reference ranges. Values outside the reference range will be flagged. Additionally, differences from baseline will be evaluated.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the RPM/DBLM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### 7.8.3 Vital signs

The analyses of vital signs will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### **7.8.4** ECG

#### 12-lead ECG

Abnormal findings will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator.

All evaluation of ECG data except of exposure response analysis will be based on the TS. The exposure-response analysis will then be done on the ECGPCS.

#### Listing of individual data

For all quantitative endpoints, listings of individual data will be shown in Appendix 16.2. Occurrences of notable findings will be flagged.

For all subjects with any notable finding in quantitative ECG recordings, a separate listing will be created as end-of-text display (based on the same display template as in Appendix 16.2), and the corresponding time profiles will be shown.

Comments regarding the ECGs will be listed.

## Analysis of central tendency

Descriptive statistics (N, mean, SD, min, median, max) will be provided for the changes from baseline over time in all ECG variables.

For QTcN, QTcF, QT and HR, a repeated measurements analysis of the changes from baseline with baseline as a covariate will be performed. The model will include the fixed effects "baseline", "treatment", "time", "baseline\*time" interaction, and "treatment\*time" interaction. The covariance model for the repeated effect "time" will be unstructured (i.e. TYPE=UN or UNR); in case of convergence problems refer to Additional Section 9.2. For each dose group and each time point, the contrast of the means for "treatment-placebo" will be estimated by the difference in the corresponding adjusted means (Least Squares Means); two-sided 90% CIs based on the t-distribution will also be computed. For each of the above ECG variables, the time profiles of the mean differences to placebo in the changes from baseline and the corresponding 90% CIs will be presented in a figure.

The following SAS code can be used to fit the model:

```
PROC MIXED DATA=indata CL METHOD=REML;
CLASS subject treat time;
MODEL ECGep = treat time base treat*time base*time / DDFM=KR CL ALPHA=0.1;
REPEATED time / TYPE=UN SUBJECT=subject;
LSMEANS treat*time / DIFF CL ALPHA=0.1;
SLICE treat*time / SLICEBY=time DIFF CL ALPHA=0.1 NOF PLOT=none;
RUN;
```

For PR, QRS, RR as well as QTcB, the time profiles of mean and SD for the changes from baseline on treatment will be displayed graphically by treatment.

<u>Plasma concentrations and relationship to QTcN, QTcF, QT interval and HR change from baseline</u>

For the following analyses, all time points with available ECG endpoints, which were derived from triple ECG measurements (Days 1, 2, 14, 15, 21, 28, 29), and corresponding plasma concentrations will be included.

The changes from baseline in QTcN ( $\Delta$ QTcN) will be investigated as response variable. The placebo subjects will be included in the analysis, with zero plasma concentrations. Time points with plasma concentrations "BLQ" in subjects in active dose groups will be ignored in this analysis.

As a first step, it will be investigated if there is a potential delayed or accelerated (e.g. metabolites) effects of the drug on QTcN. A general visual impression of the PK-QT relationship is provided by overlaying time profiles of plasma concentrations and QTcN changes from baseline ( $\Delta$ QTcN). All figures will be generated for each subject (presented in Appendix 16.1.9.2 of the CTR), as well as for means per active treatment (presented in Section 15.3 of the CTR).

In case of non-linearity or if there is evidence for a delayed effect, further models will be explored that better characterise the PK/ECG relationship (effect compartment, non-linear model etc.).

If there is no non-linearity or delayed effect seen, the relationship between BI 1467335 plasma concentrations and QTcN changes from baseline will be investigated in an exploratory manner using a random coefficient model approach to estimate the QTcN change from baseline and its 90% confidence interval at the geometric mean of the  $C_{max}$  for each dose. Additionally, the estimated slope with its 90% confidence interval will be provided. The used random coefficient model is based on Garnett et al. 2016 [R17-0553] (10):

```
PROC MIXED DATA=myDATA METHOD=REML;

CLASS subject active(ref=FIRST) time;

MODEL ECGep = conc active time / NOINT CL ALPHA=0.1 ALPHAP=0.1 DDFM=KR OUTPREDM=pred;

RANDOM INT conc / TYPE=UN SUBJECT=subject;

ESTIMATE 'Pred. value at conc. xx.xx' conc xx.xx active 1 -1 / CL ALPHA=0.1;

ESTIMATE 'Slope estimate' conc 1 / CL ALPHA=0.1;

RUN;
```

Here "ECGep" is the QTcN change from baseline, "active" is a dummy 0/1 variable indicating the active treatment (1=active, 0=placebo), "conc" is the corresponding plasma concentration value of the drug, and "xx.xx" is the given concentration value (usually the value of the geometric mean  $C_{max}$  of a given dose group). The "TYPE=UN" option causes the two specified random coefficients to have a bivariate normal distribution. In case of convergence problems see Section 9.2 for possible improvements (option "TYPE=FA0(2)" may also be used as a potential solution, it requests a G matrix estimate that is constrained to be nonnegative definite). If the note "estimated G matrix is not positive definite" occurs in the SAS log file, the random slope "conc" might be removed from the "RANDOM" statement.

When the plasma concentrations are not normally distributed, the exposure-response model can be applied to log(conc) instead of the raw concentration.

For visualization, the BI 1467335 plasma concentration against the response will be plotted as well as the (fixed effect) regression line, its 90% confidence interval and the geometric mean of  $C_{max}$  for each dose. For each subject and each time point, subtract the mean value of all individual observed  $\Delta QTc$  values from the placebo group for this time point from the individual observed  $\Delta QTc$  value for this subject and time point. This results in estimates for "individual  $\Delta\Delta QTc$ " values. These estimates should only be used for plotting purposes.

All of the above described graphical and statistical analyses will be also performed for QTcF, HR and QT in place of QTcN.

### **Categorical Endpoints**

For the categorical endpoints, frequency tables will be provided.

For subjects with notable findings, the individual time courses of QTcN, QTcF, QT, HR, PR and QRS of these subjects will be presented in figures.

#### **7.8.5** Others

Physical examination findings and ophthalmological examination findings (exclusion of cataract) will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination or ophthalmological examination findings will be prepared.

# 8. REFERENCES



8 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version



#### 9. ADDITIONAL SECTIONS

#### 9.1 DETAILED DESCRIPTION OF ENDPOINTS FOR ECG

QT, PR, QRS and RR baseline and on-treatment measurements (see <u>Table 6.7: 1</u>) are included in the centralised ECG evaluation.

For each single ECG with centralised evaluation, measurements of QT, PR, QRS and preceding RR interval of four cardiac cycles will be determined and stored in the database as raw data.

QTcF, HR and QTcB will be calculated based on the derivation rules as follows:

From the four cardiac cycles of a single ECG, the HR (measured in beats/min) will be calculated as

$$HR [beats/min] = \frac{60\ 000}{\overline{RR}}$$

where  $\overline{RR}$  is the mean of the four RR intervals (measured in msec).

Similarly, the QT interval corrected for HR according to Fridericia's formula (QTcF) for a single ECG will be derived as

$$QTcF [msec] = \sqrt[3]{\frac{1000}{\overline{RR}}} \overline{QT},$$

where  $\overline{QT}$  is the mean of the four QT intervals and  $\overline{RR}$  is the mean of the corresponding preceding RR intervals of the four cardiac cycles for this ECG.

Likewise, the HR-corrected QT interval according to Bazett's formula (QTcB) for a single ECG is given by

QTcB [msec] = 
$$\sqrt[2]{\frac{1000}{\overline{RR}}}\overline{QT}$$
.

In addition, data dependent population heart rate correction QTcN will be derived for a given pair of QT and RR values as

QTcN [msec] = 
$$\left(\frac{1000}{RR}\right)^{slope} * QT[msec],$$

(RR and QT are given in msec). A common *slope* will be estimated for the whole population (all subjects in the TS) based on the random coefficient model described below. The RR and QT intervals used for this slope estimation will be the arithmetic means of the four cardiac cycles from each single ECG on baseline and on placebo. Hence, the evaluation will be based on 1098 pairs (36 subjects \* 1 central baseline ECG with triple measurement \* 3 measurements + 9 placebo subjects \* [34 central post-baseline ECGs with triple

measurement \* 3 measurements + 8 central post-baseline ECGs with single measurement]) of RR and OT interval measurements for each subject. If there is a missing baseline or placebo value, no imputed values will be used in the analysis described in the following:

A random coefficient model with covariate "log-transformed RR interval" is fit (natural log), which accounts for subject effects (Ring [R10-2920] (11)):

$$Y_{ik} = \mu_0 + s_{0k} + (\delta_1 + s_{1k})x_{ik} + \varepsilon_{ik}$$
,

where

log-transformed QT interval of the  $i^{th}$  ECG of subject k;  $Y_{ik}$ 

the overall intercept;  $\mu_0$ 

the random intercept associated with subject k; Sok

the regression effect of the covariate, i.e. the common slope associated with the  $\delta_I$ relationship between the log-transformed QT and RR intervals;

the random slope associated with subject k;  $S_{1k}$ 

 $x_{ik}$ 

log-transformed RR interval of the  $i^{th}$  ECG of subject k; the random error associated with the  $i^{th}$  ECG of subject k.  $\varepsilon_{ik}$ 

The slope is then calculated as  $\delta_1$ .

The following SAS code will be used to fit the model:

```
PROC MIXED DATA=xxxx CL METHOD=REML;
CLASS subject;
MODEL lnQT = lnRR / DDFM= KENWARDROGER ALPHA=0.05 CL;
RANDOM INT lnRR / TYPE=UN SUBJECT=subject;
ESTIMATE 'Population slope' lnRR 1 / ALPHA=0.05 CL;
RUN;
```

The PR and QRS values for a single ECG are derived as the means of the PR and QRS values, respectively, of the four cardiac cycles for this ECG.

In case of triple ECGs at a time point, the respective ECG variable will be averaged over the triple ECG measurements at this time point (arithmetic mean). Note that in case of missing values the averaging is simply done for the available values.

#### 9.2 STEPS IN CASE OF CONVERGENCE PROBLEMS FOR REPEATED **MEASURES MODEL IN ECG**

In case of convergence problems one may try one (or more) of the following steps:

- 1.) Set MAXITER=100 (or even higher for PROC GLIMMIX) and/or MAXFUNC=200 (for PROC GLIMMIX, these options are available within the NLOPTIONS statement)
- 2.) Set SINGULAR=1E-10 as option (for PROC MIXED: in the model statement)
- 3.) Use option SCORING=4 in the final run to request a Fisher scoring algorithm to be used for the first 4 iterations
- Include the additional statement in the PROC MIXED call: 4.)

PERFORMANCE NOTHREAD;

5.) Perform an initial run including the statement

ODS OUTPUT COVPARMS=covstart;

followed by a final run using

PARMS / PARMSDATA=covstart;

In the special case with the note "Convergence criteria met but final hessian is not positive definite" try instead/in addition

PARMS / OLS;

to request ordinary least squares starting values.

6.) One may also use estimates from a simpler model (e.g. using AR(1)) as starting values for the run with TYPE=UN or UNR

In case an unstructured covariance matrix (i.e. TYPE=UN or UNR) does not work, also in conjunction with all steps from 1)-6) mentioned above, the following covariance structures will be chosen, in the pre-defined order:

- Toeplitz structure with heterogeneous variances (TOEPH) for the REPEATED effect
- heterogeneous first-order autoregressive structure (ARH(1)) for the REPEATED effect
- TOEPH for both the RANDOM and the REPEATED effect
- ARH(1) for both the RANDOM and the REPEATED effect, but with the additional random statement RANDOM INT / SUBJECT=subject;

TSAP for BI Trial No: 1386.8 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 29-Aug-2017 | | None | This is the final TSAP without any |
| | | | | modification |